CLINICAL TRIAL: NCT01365208
Title: Prospective Evaluation of Plasma EBV DNA Half-life and PET-CT Scanning as a New Tool in Assessing Early Response to Chemotherapy in Patients With Advanced Nasopharyngeal Carcinoma
Brief Title: New Approach of Assessing Drug Response for Treatment of Nasopharyngeal Cancer
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Other Study IDs: NPC023
Record Dates: First submitted 2011-05-11; First posted 2011-06-03 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EBV DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- advanced nasopharyngeal carcinoma
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — platinum-based chemotherapy

SUMMARY:
The combination of pEBV DNA (half-life) and PET-CT following 1 course of chemotherapy allow earlier and more detection of drug response in advanced NPC than RECIST method, in patients with previously untreated advanced NPC who will receive platinum-based chemotherapy. This study will also determine if this new method can predict survival in these patients. This study may have far-reaching impact on drug development in NPC as it may offer a more optimal way of evaluating drug efficacy in clinical trials and also in clinical management.

ELIGIBILITY:
Inclusion Criteria:

* undergo chemotherapy for any one of the following settings:

  1. Setting 1: Neoadjuvant chemotherapy prior to cheom-RT
  2. Setting 2: Palliative chemotherapy in Chemonaive patients
  3. Setting 3: Palliative chemotherapy in previously treated patients (i.e. 2nd line or 3rd line chemo)
* Age >= 18 years
* (ECOG) performance status of 0-2
* have detectable levels of pEBV DNA at baseline
* have measurable tumor sites by RECIST criteria
* have adequate bone marrow, renal and hepatic functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: paitent with advanced nasopharyngeal carcinoma
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-07; Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
To determine if measuring tumor metabolic response during chemotherapy can predict survival | 3 years
To determine if measuring plasma EBV DNA (half-life) early during chemotherapy can predict survival | 3 years

SECONDARY OUTCOMES:
New method of assessing drug response (measuring tumor metabolic response via FDG-PET & plasma EBV DNA (half-life) after 1 course of chemotherapy) can better predict survival, than the conventional method | 3 years
To determine if plasma EBV DNA (half-life) correspond with best response rate based on the conventional 'Response Evaluation Criteria in Solid Tumors' - RECIST criteria. | 3 years
overall survival | 3 Years
progression free survival | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Ma, MD, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ma B, Hui EP, King A, Leung SF, Kam MK, Mo F, Li L, Wang K, Loong H, Wong A, Chan CM, Chan KCA, Wong SCC, Lo YMD, Chan AT. Prospective evaluation of plasma Epstein-Barr virus DNA clearance and fluorodeoxyglucose positron emission scan in assessing early response to chemotherapy in patients with advanced or recurrent nasopharyngeal carcinoma. Br J Cancer. 2018 Apr;118(8):1051-1055. doi: 10.1038/s41416-018-0026-9. Epub 2018 Mar 20. PMID 29555989